CLINICAL TRIAL: NCT02538159
Title: Randomized, Prospective, Single-center Study to Compare the Effectiveness and Safety in Terms of Catheter Bacteraemia, Between Peripherally Inserted Central Catheters and Non-tunneled Central Venous Catheter in Tertiary Hospital
Brief Title: Safety and Bacteraemia Between Peripherally Inserted and Central Inserted Catheters.
Acronym: PYCBAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-CAT-2014-36
Record Dates: First submitted 2015-04-23; First posted 2015-09-02 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Catheter Related Infections
Keywords: Non-tunneled Central venous catheter; Bacteraemia; Peripherally inserted central venous catheter
MeSH Terms: conditions — Catheter-Related Infections; Toxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental CVC (Experimental): CVC insertion Non-tunneled Central venous catheter insertion
  Interventions: Device: CVC
- Experimental PICC (Experimental): PICC insertion Peripherally inserted catheter
  Interventions: Device: PICC

INTERVENTIONS:
Device: CVC — The inclusion of any CVC is an aseptic technique, so hand washing, mask, cap is required, sterile gloves and scoping insertion using sterile drapes. The skin disinfection is carried out with 2% chlorhexidine alcohol 17, to be dried completely before insertion of the catheter (30 seconds). No prophylactic antibiotic was administered before insertion. In the case of CVC, the subclavian vein of choice will be followed by the femoral and jugular. Seldinger technique with direct radiation control in the operating room is used.
  Arms: Experimental CVC
Device: PICC — The inclusion of any PICC is an aseptic technique, so hand washing, mask, cap is required, sterile gloves and scoping insertion using sterile drapes. The skin disinfection is carried out with 2% chlorhexidine alcohol 17, to be dried completely before insertion of the catheter (30 seconds). No prophylactic antibiotic was administered before insertion. PICC vein of choice is the basilica vein with help of Ecography in the interventional radiology room.
  Arms: Experimental PICC

SUMMARY:
Clinical, prospective, single-center, national trial. open and randomized at 1: 1 to compare the rate of bacteremia associated between non-tunneled Central venous catheter and peripheral inserted central catheter.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years.
* Patients hospitalized at our institution requiring at least 6 days of intravenous treatment in a conventional ward of our hospital.
* Signed informed consent by the patient and / or when necessary parent / legal guardian.

Exclusion Criteria:

* Patients with bacteremia at the time of catheter insertion.
* Patients admitted to hematology or intensive care units, for considered a type of patient characteristics very different from other patients.
* Patients with severe clinical situation.
* Patients in whom peripheral venous access is technically impossible, patients outpatient and express refusal of the patient.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2017-06-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Bacteraemia | 30 days
  Number of participants with Bacteraemia from insertion until 30 days after remove of the catheter

SECONDARY OUTCOMES:
morbidities in catheter insertion | 1 day
  Number of participants with complications during catheter insertion
Comparison of morbidities during manipulation of the catheters | 30 days
  Number of participants with complications during manipulation of the catheters
30 days Mortality | 30 days
  Number of died participants
Visual analogic scale of Pain | 30 days
  Visual analogic scale of Pain in site of insertion from insertion until remove of the catheter
Health-care costs | 30 days
  Economic study of the whole procedure including complications

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain